CLINICAL TRIAL: NCT05039320
Title: The Effect of Oral Probiotics (Streptococcus Salivarius K12) on Biofilm, Salivation, and Secretory Immunoglobulin A Salivary Level: a Pilot Randomized Clinical Trial
Brief Title: The Effect of Probiotics on Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: I. Mechnikov Research Institute of Vaccines and Sera (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18081211
Record Dates: First submitted 2021-08-29; First posted 2021-09-09 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-08

CONDITIONS: Oral Disease
Keywords: probiotics; Streptococcus salivarius K12; dental biofilm; salivary secretory immunoglobulins A; unstimulated salivary flow rate
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - probiotic (Experimental): The use of Streptococcus salivarius K12 containing tablets ("Bactoblis", registration number: AM.01.06.01.003.Е.000024.07.18; 20.07.18, MEDICO DOMUS, d.d.o.; 18116, Nis, Serbia)) once a day for 4 weeks (before bedtime after evening brushing).
  Ingredients: basic active ingredient - Streptococcus salivarius K12 (≥1×109 CFU in 1 tablet), excipients - fructose (sweetener), maltodextrin, silicon dioxide, magnesium stearate (vegetable), strawberry flavouring.
  Interventions: Dietary Supplement: Bactoblis
- Group 2 - placebo (Placebo Comparator): The use of placebo tablets once a day for 4 weeks (before bedtime after evening brushing).
  Ingredients: fructose (sweetener), maltodextrin, silicon dioxide, magnesium stearate (vegetable), flavouring (strawberry).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bactoblis — dissolve the tablets in the mouth once a day for 4 weeks
  Other Names: Probiotic: Streptococcus salivarius K12
  Arms: Group 1 - probiotic
Dietary Supplement: Placebo — dissolve the tablets in the mouth once a day for 4 weeks
  Arms: Group 2 - placebo

SUMMARY:
This will be a double-blind, randomized, placebo-controlled two-arm parallel groups study of the effect of oral probiotics containing Streptococcus salivarius K12 on oral biofilm, salivation rate, and secretory immunoglobulin A salivary level.

The aim of the study is to assess the effect of oral probiotics containing Streptococcus salivarius K12 strain on oral biofilm, unstimulated salivary flow rate, and salivary secretory immunoglobulin A (sIgA) levels.

DETAILED DESCRIPTION:
Thirty consenting patients aged 20-24 years who will meet the inclusion criteria will be recruited in the study. At the preparatory phase patients will be recruited and randomized, their oral hygiene protocols will be standardized, researchers will be calibrated and trained. The main phase will include a double-blind, randomized, two-arm parallel group, placebo-controlled study of probiotics effects, and wash-out period. Patients will be randomly divided into 2 groups (group 1 - probiotics, group 2 - placebo). Clinical examination will be performed at baseline, after 4 weeks (probiotic/placebo intake) and 6 weeks (wash-out), and will include the assessment of DMFT index, oral hygiene level (the Turesky Modification of the Quigley-Hein Plaque Index (TMQHPI)), gingival inflammation (PMA index), salivation rate (unstimulated salivary flow), and salivary concentration of secretory immunoglobulins A.

The study is estimated to complete enrollment within 4 weeks from study initiation; however, enrollment will remain open until the study goal is met. The duration of this study for each subject will be a maximum of eight (10) weeks: 4 weeks - preparatory period, 4 weeks - intervention period, and wash out period (2 weeks).

Screening (First) visit

* Review the study with the subject and obtain written informed consent
* Assign the subject a unique screening/enrollment number
* Review and record medical history, and medication history to determine eligibility based on inclusion/exclusion criteria
* Record demographics (age, gender)
* Document vitals
* Document all current medications, including medications over-the-counter and herbal medications
* Perform physical examination

  * Determine DMFT index
  * Determine oral hygiene level (TQHPI)
* Provide training in standardised brushing techniques.

The allocation concealment will be performed by the use of containers numbered by a "third party" (person, who will not participate in the study). The tablets in the bottles without titles will be placed in the containers. The tablets in different groups will look similar. The patient on enrollment will receive a container with tablets. Neither patients nor researchers will be aware of the type of a tablets received by each patient (double blinding).

Baseline (Second) visit (4 weeks from the Screening visit) - all groups

- Perform physical examination

* Determine DMFT index
* Determine oral hygiene level (TQHPI)
* Determine gingival tissue condition (PMA index)
* Determine unstimulated salivary flow rate
* Determine a concentration of secretory immunoglobulins A in saliva (ELISA)

Third visit (4 weeks from the Baseline visit) - all groups

- Perform physical examination

* Determine DMFT index
* Determine oral hygiene level (TQHPI))
* Determine gingival tissue condition (PMA index)
* Determine unstimulated salivary flow rate
* Determine a concentration of secretory immunoglobulins A in saliva (ELISA)
* Assess for adverse events

Fourth visit (2 weeks from the Third visit) = Final Study Visit - all groups

* Perform physical examination • Determine DMFT index

  • Determine oral hygiene level (TQHPI))

  • Determine gingival tissue condition (PMA index)
  * Determine unstimulated salivary flow rate
  * Determine a concentration of secretory immunoglobulins A in saliva (ELISA)
  * Assess for adverse events

Early Termination visit

* Assess for adverse events
* Assess for complications following treatments
* Document all current medications, including medications over-the-counter and herbal medications

Preparatory phase of the study Patient training Oral hygiene instructions will be given and the compliance with the recommendations will be controlled with weekly visits to the dental office. The participants will be familiarized with the assessment techniques and trial procedures Qualification and calibration of the observers The clinical examinations will be performed by two dentists who are the members of Therapeutic Dentistry Department, Sechenov University, Moscow, Russia. The examiners will be trained and calibrated to obtain an intra- and inter-examiner agreement of 90%, using Kappa statistics.

Randomization Thirty people aged 20-24 years will be examined and randomly assigned to one of the study groups: Group 1 will use tablets containing probiotic (Streptococcus salivarius K12). Group 2 will use tablets containing placebo. The allocation concealment will be performed by the use of containers numbered by a "third party" (person, who will not participate in the study). The tablets in bottles without any titles will be placed in the containers. The tablets in both groups will look similar. The patient on enrolment will receive a container of tablets. Neither patients nor researchers will be aware of the type of tablets used.

Treatment protocol The patients will use the prescribed tablets ("Bactoblis", registration number: AM.01.06.01.003.Е.000024.07.18; 20.07.18, MEDICO DOMUS, d.d.o. (18116, Nis, Serbia)) for 4 weeks 1 tablet per day. The end of the treatment course will be followed by a two-week wash-out period. During the wash-out period, patients will have to stop taking their prescribed tablets. A wash-out period is necessary to assess the stability of the results achieved. Control examinations will be carried out in the following periods: 4 weeks and 6 weeks.

Physical examination

The examination will include determination of:

DMFT index, oral hygiene level (TQHPI), gingival tissue condition (PMA index), unstimulated salivary flow rate, and a concentration of secretory immunoglobulins A in saliva (ELISA).

Data collection and reporting. Data will be collected at the following points: at baseline, and after 4 and 6 weeks of the study.

Data from the study will be maintained for two (2) years after the date the investigation is completed, terminated or until the records are no longer required to support the protocol, whichever date is later. Patient records and data are eligible for inspection and/or copying by applicable regulatory authorities.

Data handling and record keeping Data entry will be completed in the RedCap database (which will cover all the created CRFs). The data will be exported into CSV file format, which will then be used for data analysis. Only de-identified data will be used for data analysis. All hard copy documents will be shredded within five years after completion of the study upon Sponsor approval. Collected de-identified data will be sent to a biostatistician for statistical analysis.

Adverse reactions. There is no expectation of any adverse outcomes or reactions due to a patient using probiotics or placebo. However, hypersensitivity reactions to some of the tablets' components are still possible. All participants will be given access to contact info of the investigators. Any adverse reactions should be reported immediately to the investigators.

Reasons for Withdrawal or Termination

The following is a list of possible reasons for study treatment discontinuation:

* Screening Failure
* Subject withdrawal of consent
* Subject is not compliant with study procedures
* Adverse Event that in the opinion of the Investigator would be in the best interest of the subject to discontinue study participation
* Protocol violation requiring discontinuation
* Lost to follow-up All subjects are free to withdraw from participation at any time, for any reason, specified or unspecified, and without prejudice.

Statistical analysis plan All analyses will be performed using per-protocol population: all subjects will be analyzed who did not substantially deviate from the protocol as to be determined on a per-subject basis by the study principal investigator immediately before database lock.

Data will be presented as means and standard deviations with 95% confidence intervals, medians and 25 and 75 percentiles, and percentages depending on the type of variables. The normality and sphericity of distribution of continuous variables will be assessed with Shapiro-Wilk and Leven's tests, respectively. If the assumptions of normality and sphericity are satisfied, repeated measures mixed ANOVA model will be performed followed by post-hoc Tukey test with adjustment for multiple comparisons. If the aforementioned assumptions are not satisfied, the differences between groups will be assessed using Mann-Witney U-test and the difference within the groups at different study timepoints will be assessed with Friedman test with post-hoc comparisons. The same non-parametric tests will be used for the analyses of categorical and ordinal variables. Fisher's exact test will be used to access the frequencies of categorical variables in the groups. Correlation between Salivation rate, salivary sIgA concentration, TQHPI, DMFT, Decay, and PMA will be assessed using Spearman correlation coefficient.

All summary tables will be structured with a column for each timepoint and rows for each assessed outcome and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

ELIGIBILITY:
Inclusion Criteria:

* Permanent bite;
* Presence of more than 20 teeth;
* Absence of systemic and chronic diseases.

Non-inclusion Criteria:

* More than 5 cavities requiring treatment;
* Refusal to sign informed consent;
* Taking supplements and medication containing probiotics or prebiotics 3 weeks before the study;
* Taking antibiotics (within 1 month before the study);
* Orthodontic and prosthetic treatment;
* Allergy to the components of the drugs used in the study.

Exclusion Criteria:

* Use of other hygiene products, immunostimulants and antibacterials, probiotics, prebiotics during the study;
* Refusal to take a given medication;
* Failure to attend check-ups.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Changes in the concentration of secretory immunoglobulin A in saliva | 4 weeks after the baseline
  Salivary secretory IgA levels are determined using the 8668 IgA secretory ELISA-BEST kit (VectorBest, Novosibirsk, Russia) based on a two-step "sandwich" version of the enzyme-linked immunosorbent assay (ELISA).
Changes in the concentration of secretory immunoglobulin A in saliva | 6 weeks after the baseline
  Salivary secretory IgA levels are determined using the 8668 IgA secretory ELISA-BEST kit (VectorBest, Novosibirsk, Russia) based on a two-step "sandwich" version of the enzyme-linked immunosorbent assay (ELISA).
Changes in the unstimulated salivary flow rate | 4 weeks after the baseline
  participants refrain from eating, drinking, smoking, or conducting oral hygiene for a minimum of 90 minutes prior to salivary collection. To avoid diurnal variations in saliva output, all measurements are taken in the morning. Participants are comfortably seated and, after a few minutes of relaxation, are trained to avoid swallowing saliva and asked to lean forward and spit all the saliva they produce every 2 minutes through a glass funnel and into a graduated test tube. The volume collected for 10 minutes is measured. The flow rate is determined according to the formula: Salivation rate(ml/min) = saliva volume(ml) / saliva collection time(min).
Changes in the unstimulated salivary flow rate | 6 weeks after the baseline
  participants refrain from eating, drinking, smoking, or conducting oral hygiene for a minimum of 90 minutes prior to salivary collection. To avoid diurnal variations in saliva output, all measurements are taken in the morning. Participants are comfortably seated and, after a few minutes of relaxation, are trained to avoid swallowing saliva and asked to lean forward and spit all the saliva they produce every 2 minutes through a glass funnel and into a graduated test tube. The volume collected for 10 minutes is measured. The flow rate is determined according to the formula: Salivation rate(ml/min) = saliva volume(ml) / saliva collection time(min).

SECONDARY OUTCOMES:
Turesky Modification of the Quigley-Hein Plaque Index | 4 weeks after the baseline
  A plaque detection solution is used to detect the presence of plaque on both the vestibular and oral surfaces of all teeth except the third molars. Each surface is divided into 3 segments: mesial, central and distal. Thus, 6 segments are evaluated for each tooth.
  Evaluation criteria:
  0 - no staining;
  1. - separate areas of plaque in the cervical part;
  2. - plaque in the form of a thin continuous band up to 1 mm wide in the cervical part;
  3. - cervical part is covered by plaque that is more than 1 mm wide, but less than 1/3 of the tooth crown;
  4. - plaque covers 1/3 to 2/3 of the crown;
  5. - plaque covers more than 2/3 of the crown.
Turesky Modification of the Quigley-Hein Plaque Index | 6 weeks after the baseline
  A plaque detection solution is used to detect the presence of plaque on both the vestibular and oral surfaces of all teeth except the third molars. Each surface is divided into 3 segments: mesial, central and distal. Thus, 6 segments are evaluated for each tooth.
  Evaluation criteria:
  0 - no staining;
  1. - separate areas of plaque in the cervical part;
  2. - plaque in the form of a thin continuous band up to 1 mm wide in the cervical part;
  3. - cervical part is covered by plaque that is more than 1 mm wide, but less than 1/3 of the tooth crown;
  4. - plaque covers 1/3 to 2/3 of the crown;
  5. - plaque covers more than 2/3 of the crown.
Papillary-marginal-alveolar index | 4 weeks after the baseline
  The test is assessed by applying iodine-containing solution to the gingiva around all teeth. The test is negative if the mucosa has a light yellow color. In the presence of gingival inflammation, a yellow-brown staining of varying intensity is observed. The PMA index is assigned to each gingival unit of the maxillary and mandibular teeth as follows: 0, no inflammation and 1, inflammation. The total PMA index score is calculated for each patient accordingly. This index evaluates the number of gingival units (papillary, marginal, and attached gingiva) exhibiting gingival inflammation around erupted teeth.
Papillary-marginal-alveolar index | 6 weeks after the baseline
  The test is assessed by applying iodine-containing solution to the gingiva around all teeth. The test is negative if the mucosa has a light yellow color. In the presence of gingival inflammation, a yellow-brown staining of varying intensity is observed. The PMA index is assigned to each gingival unit of the maxillary and mandibular teeth as follows: 0, no inflammation and 1, inflammation. The total PMA index score is calculated for each patient accordingly. This index evaluates the number of gingival units (papillary, marginal, and attached gingiva) exhibiting gingival inflammation around erupted teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Ksenia Babina, PhD, Study Director — Sechenov University
Locations (1):
- Institute of Dentistry of Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polyakova MA, Arakelyan MG, Babina KS, Margaryan EG, Sokhova IA, Doroshina VY, Novozhilova NE. Qualitative and Quantitative Assessment of Remineralizing Effect of Prophylactic Toothpaste Promoting Brushite Formation: A Randomized Clinical Trial. J Int Soc Prev Community Dent. 2020 May 7;10(3):359-367. doi: 10.4103/jispcd.JISPCD_493_19. eCollection 2020 May-Jun. PMID 32802784
- [Derived] Babina K, Salikhova D, Polyakova M, Svitich O, Samoylikov R, Ahmad El-Abed S, Zaytsev A, Novozhilova N. The Effect of Oral Probiotics (Streptococcus Salivarius k12) on the Salivary Level of Secretory Immunoglobulin A, Salivation Rate, and Oral Biofilm: A Pilot Randomized Clinical Trial. Nutrients. 2022 Mar 7;14(5):1124. doi: 10.3390/nu14051124. PMID 35268099